CLINICAL TRIAL: NCT04934462
Title: Prospective Evaluation of Non-Surgical and Arthroscopic Treatment for Hip Microinstability
Brief Title: Evaluation of Non-Surgical and Arthroscopic Treatment for Hip Microinstability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Society of Medicine (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hip Microinstability Study
Record Dates: First submitted 2021-05-31; First posted 2021-06-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Musculoskeletal Abnormalities; Hip Injuries
Keywords: arthroscopy; physiotherapy
MeSH Terms: conditions — Musculoskeletal Abnormalities; Hip Injuries | interventions — Physical Therapy Modalities; Arthroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-surgical treatment (Other): All participants will undergo 6 months of non-surgical treatment.
  Interventions: Procedure: physiotherapy
- arthroscopic treatment (Other): Those participants with failed non-surgical treatment at 6 months will undergo arthroscopic treatment.
  Interventions: Procedure: physiotherapy; Procedure: arthroscopy

INTERVENTIONS:
Procedure: physiotherapy — Six months physiotherapy aimed at hip stability.
Procedure: arthroscopy — Arthroscopic plication of hip joint capsule.
  Arms: arthroscopic treatment

SUMMARY:
Microinstability of the hip joint is an important cause of hip pain and reduced hip function in young and active individuals. Hip microinstability is due to extraphysiologic hip motion and could be secondary to acetabular dysplasia, connective tissue disorder, macrotrauma, microtrauma, iatrogenic- and idiopathic causes. Treatment for hip microinstability is initiated with non-surgical treatment consisting of physiotherapy aimed mainly at stability. If non-surgical treatment fails, surgery with arthroscopic plication of the hip joint capsule is the preferred method. This study evaluates non-surgical and arthroscopic treatment for hip microinstability regarding hip function and adverse events.

DETAILED DESCRIPTION:
This is a prospective cohort study evaluating 26 participants above 18 years of age undergoing non-surgical and surgical treatment for microinstability of the hip joint. Participants with findings on physical examination and imaging suggestive of hip microinstability will undergo six months of physiotherapy aimed at stabilizing the hip joint. If non-surgical treatment fails, a diagnostic hip arthroscopy will be performed, and if hip microinstability is confirmed, the participants will undergo a plication of the hip joint capsule. Participants will be evaluated with Patient-Reported Outcome Scores (PROMs) and strength- and function tests at time of enrollment and at 6-, 12- and 24 months following treatment. The primary outcome is hip function determined by PROMs and strength- and function tests. Secondary outcomes include Health-Related Quality of Life (HRQL), sport activity level and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Hip microinstability
* Minimum 18 years old

Exclusion Criteria:

* Hip osteoarthritis
* Severe hip dysplasia
* Perthes disease or avascular necrosis of the femoral head
* Previous surgery to the hip joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Hip Function on the International Hip Outcome Tool (iHOT-12) at 24 Months | 24 Months
  Participant-reported hip function. Minimum score 0, maximum score 100 (higher score mean a better outcome).
Mean Change from Baseline in Hip Function on the Copenhagen Hip and Groin Outcome Score (HAGOS) at 24 Months | 24 Months
  Participant-reported hip function. Minimum score 0, maximum score 100 (higher score mean a better outcome).
Mean Change from Baseline in Maximal Isometric Hip Muscle Force in Newton at 24 Months | 24 Months
  Maximal hip isometric muscle force will be assessed using a dynamometer (Hoggan MicroFET2, Hoggan, Scientific L.L.C., Salt Lake City, USA) for hip flexion, adduction, abduction, and extension. The maximal developed force in Newton will be recorded. Higher Newton value means a better outcome.
Mean Change from Baseline in Hop Performance at 24 Months | 24 Months
  Hop performance will be measured with 3 single-leg hops: vertical hop (Muscle lab, Ergotest Technology, Oslo, Norway), hop for distance and a 30-second side-hop test. Each hop test is performed with the patients holding their hands behind their back. For the vertical hop, the time from take-off to landing is converted into hop height in centimeters. In the hop for distance test, the distance between top of the toes at take-off to heel at landing is measured in centimeters. For the 30 second side hop test, one trial per leg is allowed, where the patient is instructed to hop as many times as possible over 2 lines 40 centimeters apart. The number of hops is recorded. Higher height, longer distance and higher number of hops means a better outcome.

SECONDARY OUTCOMES:
Mean Change from Baseline in Hip Function on the EuroQoL-5 Dimensions (EQ-5D) at 24 Months | 24 Months
  Participant-reported health-related quality of life. Minimum score 0, maximum score 1 (higher score mean a higher health-related quality of life).
Mean Change from Baseline in Hip Function on the Hip Sport Activity Scale (HSAS) at 24 Months | 24 Months
  Participant-reported sport activity level. Minimum score 0, maximum score 8 (higher score mean a higher sport activity level).
Type and Number of Adverse Events at 24 Months | 24 Months
  Adverse events collected via phone interview.
Single Question "Satisfied with Treatment?" at 24 Months | 24 Months
  Participant-reported satisfaction with treatment (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Sansone, MD, PhD, Study Director — Göteborg University
Locations (3):
- Sweden (3):
  - GHP Ortho Center Göteborg, Gothenburg
  - University of Gothenburg, Gothenburg
  - Capio Artro Clinic, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ohlin A, Senorski EH, Sansone M, Leff G, Desai N, Lindman I, Ayeni OR, Safran MR. Protocol for a multicenter prospective cohort study evaluating arthroscopic and non-surgical treatment for microinstability of the hip joint. BMC Musculoskelet Disord. 2022 Mar 31;23(1):309. doi: 10.1186/s12891-022-05269-x. PMID 35361185